CLINICAL TRIAL: NCT00766272
Title: Gait Rehabilitation for Multiple Sclerosis Using Robot-assisted Body-weight-supported Treadmill Training (Lokomat)
Brief Title: Lokomat Training Effects on MS Gait Abnormalities
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study re-designed
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LO-0003
Record Dates: First submitted 2008-10-02; First posted 2008-10-03 (Estimated); Last update posted 2013-09-23 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis
Keywords: Rehabilitation; Treadmill; MS; Gait; Robot
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Body-weight supported treadmill training
  Interventions: Device: Lokomat

INTERVENTIONS:
Device: Lokomat — Body-weight will be supported using a harness, which suspends the subject above a motorized treadmill (Lokomat, Hocoma, Zurich, Switzerland). The system also incorporates a robot-driven gait orthotic, called the Lokomat, which will be secured to the subject's lower extremity and pelvis using adjustable cuffs and pads. The Lokomat uses computer-controlled motors to drive the hips and knees toward more normative kinematic patterns for gait.

SUMMARY:
Multiple sclerosis is a degenerative disease that affects more than 400,000 people in the US alone. MS is in fact the most common disabling neurological disorder in young adults. Symptoms of the disease can include problems with balance, walking, fatigue, weakness and vision. Over 85% of people with Multiple Sclerosis have problems walking. This can cause them to fall or have a constant fear of falling. To prevent falling, MS patients rely on equipment, such as walkers and canes. These costs can cause financial difficulties for MS patients and families.

A significant problem that is only recently being studied is the relationship between falling and MS. Recent studies have shown that MS patients fall more often than those without MS, and also fall more than the elderly population. The consequent fear of falling is also an important problem, as those worried about falling will probably change their daily habits to lower their risk. This can mean keeping from certain physical and social activities or even staying indoors. Thus, falls and fear of falling can have negative medical, physical, psychological, and social consequences for the patient.

Improving patients' walking may help reduce falls and the fear of falling. Treadmill training has been shown to improve walking in patients with MS and to lower their risk of falling. One way to train patients on a treadmill is with the use of robots that can help move their limbs in a more normal way. This kind of robot-assisted treadmill training may provide even greater benefits than treadmill training alone.

The study is expected to last 6-7.5 months. One group of participants will receive weekly telephone calls and will be asked questions on other physical activities, falls, and activity limitations the patient had during the week. Participants assigned to robot-assisted treadmill training will receive twice weekly training session for 8 weeks, for a total of 16 sessions. Each session will last about 65 to 90 minutes.

The goal of this study is to see if robot-assisted treadmill training will reduce falls and fear of falling in patients with MS. Robot-assisted treadmill training has been shown to be effective in reducing falls and fear of falling in Parkinson's disease patients. This type of training has not been tested in patients with Multiple Sclerosis. The proposed study will help to address this gap and also provide additional data on other possible improvements due to robot-assisted treadmill training including ambulation, social participation, fatigue, and balance.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS by McDonald criteria
2. Ability to clearly understand written and oral direction in English
3. Self-reported gait problem
4. One or more falls in the past 6 months
5. The ability to walk 25 feet with no more than a cane for assistance (The subject must be comfortable using a cane)
6. Age 18-70
7. Written informed consent to participate in the study
8. Approval from subject's primary care physician for physical activity

Exclusion Criteria:

1. No relapse within the last 3 months
2. No more than two relapses within the past 12 months
3. Recent myocardial infarction
4. Uncontrolled hypertension or diabetes
5. Symptomatic fall in blood pressure when standing
6. Vascular claudication or pitting edema
7. Cognitive impairments that limit comprehension of protocol instructions (assessed by Comprehension Test of Consent Form)
8. Body weight over 150 kg
9. FES-I < 25
10. Lower extremity injuries that limit range of motion or function
11. Joint problems (hip or leg) that limit range of motion or cause pain with movement
12. Unstable fractures
13. Pressure sores with any skin breakdown in areas in contact with the body harness or the robot-driven gait orthotic apparatus
14. Currently enrolled in an alcohol or drug treatment program
15. A complicating medical condition that would prevent completion of the trial
16. Enrolled in or planning to enroll in another interventional research trial using procedures proposed to enhance or limit the function of the upper or lower extremities (such as adjuvant rehabilitation or Botox injections) during the 24 weeks of participation
17. A difference of more than 2cm between subjects' right and left leg lengths
18. Unable to be properly fit into the harness or Lokomat device
19. Hypertonicity or spasticity that it interferes with a proper fit into the Lokomat
20. Pregnancy at enrollment, as determined by a home pregnancy test kit at screening visit

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Frequency of Falls | 6-7.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Albert Lo, MD PhD, Principal Investigator — Providence VA Medical Center
Locations (1):
- Providence VA Medical Center, Providence, Rhode Island, United States